CLINICAL TRIAL: NCT02576496
Title: A Phase 1 Trial to Investigate the Safety, Pharmacokinetic Profiles and the Efficacy of Tinostamustine, a First-in-Class Alkylating Histone Deacetylase Inhibition (HDACi) Fusion Molecule, in Relapsed/Refractory Hematologic Malignancies
Brief Title: Study of Tinostamustine, First-in-Class Alkylating HDACi Fusion Molecule, in Relapsed/Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDO-S101-1001
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Hematological Malignancies; Multiple Myeloma; Hodgkin's Lymphoma; Cutaneous T Cell Lymphoma
Keywords: phase 1 clinical trial; multiple myeloma; Hodgkin's lymphoma; cutaneous T-cell lymphoma; tinostamustine
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous | interventions — tinostamustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (15):
- Tinostamustine 20mg/m2 over 60min (Experimental): Tinostamustine as a single agent administered by IV infusion on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine
- Tinostamustine 40mg/m2 over 60min (Experimental): Tinostamustine as a single agent administered by IV infusion on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine
- Tinostamustine 60mg/m2 over 60min (Experimental): Tinostamustine as a single agent administered by IV infusion on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine
- Tinostamustine 80mg/m2 over 60min (Experimental): Tinostamustine as a single agent administered by IV infusion on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine
- Tinostamustine 100mg/m2 over 60min (Experimental): Tinostamustine as a single agent administered by IV infusion on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine
- Tinostamustine 120mg/m2 over 60min (Experimental): Tinostamustine as a single agent administered by IV infusion on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine
- Tinostamustine 80mg/m2 over 45min (Experimental): Tinostamustine as a single agent administered by IV infusion on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine
- Tinostamustine 60mg/m2 over 30min (Experimental): Tinostamustine as a single agent administered by IV infusion on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine
- Tinostamustine 80mg/m2 over 30min (Experimental): Tinostamustine as a single agent administered by IV infusion on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine
- Stage 2 cohort 1: relapsed/refractory Multiple Myeloma (Experimental): Tinostamustine as a single agent administered at a dose of 60mg/m2 by IV infusion over 60min on D1 and D15 of 28-day cycle.
  Interventions: Drug: Tinostamustine
- Stage 2 cohort 2: relapsed/refractory Hodgkin Lymphoma (Experimental): Tinostamustine as a single agent administered at a dose of 100mg/m2 by IV infusion over 60min on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine
- Stage 2 cohort 3: relapsed/refractory peripheral T-cell lymphoma (PTCL) (Experimental): Tinostamustine as a single agent administered at a dose of 100mg/m2 by IV infusion over 60min on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine
- Stage 2 cohort 4: relapsed/refractorycutaneous T-cell lymphoma (CTCL) (Experimental): Tinostamustine as a single agent administered at a dose of 100mg/m2 by IV infusion over 60min on D1 of 21-day cycle. Patients are of subtypes mycosis fungoides (MF) or Sézary syndrome (SS).
  Interventions: Drug: Tinostamustine
- Stage 2 cohort 5: relapsed/refractory T-cell Prolymphocytic leukemia (T-PLL) (Experimental): Tinostamustine as a single agent administered at a dose of 100mg/m2 by IV infusion over 60min on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine
- Substudy (Experimental): Tinostamustine as a single agent administered at a dose of 100mg/m2 by IV infusion over 100min on D1 of 21-day cycle.
  Interventions: Drug: Tinostamustine

INTERVENTIONS:
Drug: Tinostamustine
  Other Names: EDO-S101

SUMMARY:
This study evaluates the efficacy, safety and pharmacokinetics of tinostamustine (EDO-S101) in patients with relapsed/refractory hematologic malignancies. All patients will receive tinostamustine.

DETAILED DESCRIPTION:
Tinostamustine is a First-in-Class Alkylating Histone Deacetylase Inhibition (HDACi) Fusion Molecule. It is anticipated that tinostamustine may have activity in various hematological malignancies and solid tumors.

This study is a multi-centre, open-label phase 1 study of single agent EDO-S101 in subjects with relapsed/refractory haematological malignancies and for whom no other therapies are available.

The study consists of 2 stages and 1 sub-study:

* Stage 1: Dose Escalation to determine Maximum Tolerated Dose (MTD) at the optimal infusion time and the pharmacokinetic (PK) profiles; is expected to enroll between 21 and 48 patients. Stage 1 has now been completed.
* Stage 2: Expansion in five Cohorts, in which approximately 12-16 patients will be enrolled per cohort, for a maximum of 70 patients.

In Stage 1, tinostamustine doses were escalated following the standard 3+3 design. The decision to escalate to the next dose level occurred after all cohort patients completed 3 weeks (21 days) of observation and have been evaluated for safety and toxicity. The starting dose was a 1 hour infusion of 20 mg/m2, and the maximum dose level was 150 mg/m2. Reduced infusion times of 45 minutes and 30 minutes were assessed once the maximum tolerated dose at a 1-hour infusion was determined.

In Stage 2, five cohorts of patients (with relapsed/refractory multiple myeloma (MM); relapsed/refractory Hodgkin's lymphoma; relapsed/refractory peripheral T-cell lymphoma (PTCL); relapsed/refractory cutaneous T-cell lymphoma (CTCL); and relapsed/refractory T-cell Prolymphocytic leukemia (T-PLL) will be enrolled and treated at the recommended Phase 2 dose (RP2D) based on results of Stage 1. For MM patients, treatment will occur on Day 1 and Day 15 of a 28 day cycle. For lymphoma patients, treatment will occur on Day 1 of a 21 day cycle. Patients in each stage of the study are expected to receive a median of four Cycles of therapy, and the maximum number of treatment Cycles allowed is 12.

A sub study portion was added to the protocol as an amendment. In the sub study 6-12 patients will be treated with 100mg/m2 tinostamustine infusion delivered over 100 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient willing and able to sign an informed consent.
2. Patients age ≥18 years at signing the informed consent.
3. Life expectancy > 3 months.
4. Diagnosis of relapsed or refractory lymphoid malignancy for which there are no available therapies.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤2
6. Absolute Neutrophil Count >1,000 µL
7. Platelets ≥100,000 µL
8. Aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≤2.5 upper limit of normal (ULN).
9. Total bilirubin <2.0 mg/dL unless elevated due to known Gilbert's syndrome.
10. Creatinine ≤1.5 x ULN.
11. Serum potassium and magnesium at least at the lowest limit of normal (LLN) at baseline(before every IMP administration; if it is below LNN, (supplementation is permissible).
12. Males and females of child-bearing potential, and their partners, must be willing to use at least two effective forms of birth control during the study drug administration and for at least 90 days after the administration of the study drug to be eligible to participate. Vasectomized partners and patients must be willing to use a secondary method of effective birth control. Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient.

Specific Eligibility Criteria for Each Patient Cohort in Stage 2 Phase of the Study

Cohort 1: relapsed/refractory multiple myeloma (Recruitment to this cohort stopped Dec 2021) 1. At least one line of prior systemic therapy and no other standard therapy available with proven clinical benefit.

Cohort 2: relapsed/refractory Hodgkin's lymphoma

1. At least two lines of prior therapy and no other standard therapy available with proven clinical benefit.

Cohort 3: PTCL (recruitment to this cohort stopped March 2021)

1. Only PTCL patients with histologically or cytologically confirmed Peripheral T-Cell Lymphoma - Not Otherwise Specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), or Anaplastic Large Cell Lymphoma (ALCL).
2. At least one line of prior combination therapy and no other standard therapy available with proven clinical benefit

Cohort 4: relapsed/refractory cutaneous T-cell lymphoma (CTCL), subtypes mycosis fungoides (MF) and Sézary syndrome (SS)

1. Only CTCL patients with histologically or cytologically confirmed MF or SS with stage IIb to IVb disease based on modified ISCL/EORTC staging.
2. At least one line and a maximum of four prior standard systemic therapies and no other standard therapy available with proven clinical benefit.

Cohort 5: PTCL (Recruitment to this cohort stopped March 2021)

Eligibility criteria for sub study:

Diagnosis of relapsed or refractory lymphoma, including Diffuse large B cell lymphoma who failed at least 2 lines of prior systemic therapy, Hodgkin lymphoma who failed at least 3 lines of prior systemic therapy, follicular lymphoma grade 1-3a, marginal zone lymphoma and mantle cell lymphoma who failed at least 2 lines of prior systemic lines of prior therapy, T cell lymphoma (including PTCL, CTCL) who failed at least 2 lines of prior systemic therapy for which there are no available therapies. Patients with bulky disease and Multiple Myeloma patients are excluded from this sub study.

Exclusion Criteria:

1. Patients with any central nervous system involvement.
2. Patient who had a hematologic malignancy that has transformed.
3. Any patient who has relapsed within 100 days of stem cell infusion following an allogenic or an autologous bone marrow transplant.
4. Patients with corrected QT (QTc) interval (Fridericia's formula) > 450 msec.
5. Patients who are on treatment with drugs known to prolong the QT/QTc interval.
6. Any serious medical condition that interferes with adherence to study procedures.
7. Patients with a history of another malignancy diagnosed within three years of study enrollment excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
8. Pregnant or breast feeding females.
9. New York Heart Association (NYHA) stage III/IV congestive heart failure. The following arrhythmias not adequately controlled, active: atrial fibrillation/flutter with poor rate control, documented sustained ventricular tachycardia (defined as >30 seconds or requiring cardioversion before 30 seconds have elapsed) or TdP.
10. Active infections, or other significant co-morbidities [(e.g., active central nervous system metastases and/or carcinomatous meningitis, active infection requiring systemic therapy, history of human immunodeficiency virus (HIV) infection, or active Hepatitis B or Hepatitis C.
11. Previous cancer therapies within three (3) weeks of dosing as long as the patient has recovered to eligibility levels prior to treatment in this study.
12. Use of other investigational agents within 30 days or 5 half-lives prior to the first dose of study drug unless patient has recovered from any related toxicities ≥ Grade 1.
13. Steroid treatment within seven (7) days prior to study treatment. Patients that require intermittent use of bronchodilators, topical steroids or local steroid injections will not be excluded from the study. Patients who have been stabilized to 10 mg PO QD or less seven (7) days prior to study drug administration are allowed.
14. Patients on Valproic Acid for any indication (epilepsy, mood disorder) must be excluded from the trial .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 10-20 months from beginning of stage 2
  Determine overall response rate
Clinical benefit rate by cohort | 10-20 months from beginning of stage 2
  Determine clinical benefit rate by cohort

SECONDARY OUTCOMES:
Time to objective response | 10-20 months after beginning stage 2
  Evaluate time to objective response by cohort
Duration of response | 10-20 months after beginning stage 2
  Evaluate duration of response
Progression free survival (PFS) | 32-36 months after beginning stage 2
  Determine time to progression free survival time for patients who received the RP2D
Overall Survival (OS) | 32-36 months after beginning stage 2
  Determine the overall survival time for patients who received the RP2D

CONTACTS AND LOCATIONS:
Overall Officials: Pier L Zinzani, MD,PhD, Principal Investigator — University of Bologna Medical Center, Bologna
Locations (18):
- United States (4):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Columbia University Medical Center, New York, New York
  - University Hospitals Cleveland Seidman Cancer Center, Cleveland, Ohio
- France (5):
  - CHU de Caen, Caen
  - CHU ESTAING Service de thérapie Cellulaire et hématologique Clinique, Clermont-Ferrand
  - CHU Lille Service des Maladies du Sang, Lille
  - Hopital Haut Leveque, Pessac
  - Centre hospitalier Lyon Sud, Pierre-Bénite
- University Hospital of Ulm, Department of Internal Medicine III, Ulm, Germany
- Italy (2):
  - Institute of Hematology "L. A. Seràgnoli", University of Bologna, Bologna
  - National Cancer Institute, Fondazione 'G. Pascale', Naples
- Netherlands (2):
  - VU medisch centrum, Amsterdam
  - Erasmus MC, Rotterdam
- Spain (3):
  - Institut Català d'Oncologia de Barcelona, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
- Kantonsspital St.Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Relevant patient listing data of de-identified patients may be reviewed
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available on request through Enquiries@napp.co.uk
Access Criteria: Available on request through Enquiries@napp.co.uk

REFERENCES:
- [Derived] Sureda A, Pinto A, Ghesquieres H, Morschhauser F, Tournilhac O, Mutsaers P, Zijlstra JM, De Filippi R, Hilgier K, Manamley N, Janik T, Zinzani PL. Safety and Efficacy of Tinostamustine in a Subpopulation of Patients With Relapsed/Refractory Hodgkin Lymphoma From a Phase I Trial. Hematol Oncol. 2025 Jan;43(1):e70000. doi: 10.1002/hon.70000. PMID 39617826